CLINICAL TRIAL: NCT03392948
Title: PERcutaneouS Coronary intErventions in Patients Treated With Oral Anticoagulant Therapy
Acronym: PERSEO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Italian Society of Invasive Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: 25/10/2017
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Acute Myocardial Infarction; Unstable Angina; Chronic Stable Angina
Keywords: atrial fibrillation; prosthetic valves; pulmonary embolism; venous thrombosis; percutaneous coronary interventions; chronic anticoagulant treatment
MeSH Terms: conditions — Angina, Unstable; Angina, Stable; Atrial Fibrillation; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 5 to 8% of patients undergoing percutaneous coronary interventions requires chronic anticoagulant therapy due to atrial fibrillation or other clinical entities. There are many possible different combinations of the antithrombotic therapy after stent implantation in these patients.

Aim of this observational study is to evaluate the real world antithrombotic treatment in patients requiring anticoagulant therapy undergoing stent implantation and to compare the clinical outcome of patients treated with new oral anticoagulant drugs compared to warfarin.

The study is prospective, performed in different Italian hospitals and aimed to enroll 1080 patients with a 1 year follow up

DETAILED DESCRIPTION:
Approximately 5 to 8% of patients undergoing percutaneous coronary interventions requires chronic anticoagulant therapy due to atrial fibrillation or other clinical entities. These patients pose particular problems when undergo percutaneous coronary intervention with stent implantation (PCI-S), because of the different antithrombotic and oral anticoagulant (OAC) strategies required after the procedure when dual antiplatelet therapy is recommended. Consequently, this scenario requires careful consideration balancing bleeding, stroke and acute coronary syndrome risks.

New oral anticoagulants (NOAC) have been compared to warfarin for stroke prevention in the setting of atrial fibrillation and all these drugs showed a similar or improved efficacy over warfarin in term of ischemic events as well as bleeding complications reduction. In particular, an important safety issue is the reduction of intracranial bleeding compared to warfarin. Currently, four different NOAC have been approved for the treatment of patients with atrial fibrillation: apixaban, edoxaban, rivaroxaban and dabigatran. The first three drugs are anti Xa inhibitors whereas the last one is a direct thrombin inhibitor.

Data regarding the combination of NOAC and antiplatelet therapy after PCI-S in patients requiring chronic anticoagulant therapy are currently scarce.

The aim of our study is to perform a prospective, multicenter, observational, controlled study on patients requiring chronic anticoagulant treatment with either vitamin K antagonists or NOAC undergoing PCI-S for concomitant coronary disease.

The primary objectives of the study are:

1. To describe the contemporary antithrombotic management during and post PCI-S in patients treated with oral anticoagulant therapy
2. To evaluate, in this context, the efficacy and safety of the different NAOC compared to warfarin regimens.

According to the observational design of the study, anticoagulant therapy (vitamin antagonists or new oral anticoagulant drugs), other pharmacological therapy as well as procedural device utilized, before, during the procedure and at follow-up will be left to the physician decision.

The events will be adjudicated by a clinical event committee (CEC) comprised of qualified physicians. The CEC is responsible for adjudicating all potential endpoint events, including death, bleeding, myocardial infarction, stent thrombosis, stroke, and coronary revascularization

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing percutaneous coronary interventions with stent and an indication for chronic anticoagulant therapy.

Exclusion Criteria:

* Patients of age < 18 years old
* Lack of written informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic disease requiring oral anticoagulant therapy (atrial fibrillation, prosthetic valves, previous pulmonary embolism, venous thrombosis) undergoing either elective, urgent or emergency percutaneous coronary interventions with stent implantation for acute or chronic coronary disease.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Event | 1 year
  major bleeding, myocardial infarction, death, stroke, myocardial revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, Principal Investigator — Ospedale Sandro Pertini, ASL RM2, Rome
Locations (10):
- Italy (10):
  - Ospedale Maggiore Carlo Alberto Pizzardi, Bologna, BO
  - Azienda Ospedaliero - Universitaria "Mater Domini", Catanzaro, CZ
  - Ospedale della Misericordia, Grosseto, GR
  - A.O.U. Policlinico "G.Martino" - Messina, Messina, ME
  - Ospedale Civile SS Annunziata, Sassari, SS
  - Ospedale SS Filippo e Nicola, Avezzano
  - Ospedale "Vito Fazzi", Lecce
  - Ospedale "Infermi" di Rimini, Rimini
  - Ospedale S. Eugenio, Roma
  - Ospedale Sandro Pertini, Roma

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make Individual Participant Data available

REFERENCES:
- [Background] Rubboli A, Colletta M, Herzfeld J, Sangiorgio P, Di Pasquale G. Periprocedural and medium-term antithrombotic strategies in patients with an indication for long-term anticoagulation undergoing coronary angiography and intervention. Coron Artery Dis. 2007 May;18(3):193-9. doi: 10.1097/MCA.0b013e328012a964. PMID 17429293
- [Background] Wang TY, Robinson LA, Ou FS, Roe MT, Ohman EM, Gibler WB, Smith SC Jr, Peterson ED, Becker RC. Discharge antithrombotic strategies among patients with acute coronary syndrome previously on warfarin anticoagulation: physician practice in the CRUSADE registry. Am Heart J. 2008 Feb;155(2):361-8. doi: 10.1016/j.ahj.2007.09.003. Epub 2007 Oct 25. PMID 18215609
- [Background] Leon MB, Baim DS, Popma JJ, Gordon PC, Cutlip DE, Ho KK, Giambartolomei A, Diver DJ, Lasorda DM, Williams DO, Pocock SJ, Kuntz RE. A clinical trial comparing three antithrombotic-drug regimens after coronary-artery stenting. Stent Anticoagulation Restenosis Study Investigators. N Engl J Med. 1998 Dec 3;339(23):1665-71. doi: 10.1056/NEJM199812033392303. PMID 9834303
- [Background] ACTIVE Writing Group of the ACTIVE Investigators; Connolly S, Pogue J, Hart R, Pfeffer M, Hohnloser S, Chrolavicius S, Pfeffer M, Hohnloser S, Yusuf S. Clopidogrel plus aspirin versus oral anticoagulation for atrial fibrillation in the Atrial fibrillation Clopidogrel Trial with Irbesartan for prevention of Vascular Events (ACTIVE W): a randomised controlled trial. Lancet. 2006 Jun 10;367(9526):1903-12. doi: 10.1016/S0140-6736(06)68845-4. PMID 16765759
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Oldgren J, Wallentin L, Alexander JH, James S, Jonelid B, Steg G, Sundstrom J. New oral anticoagulants in addition to single or dual antiplatelet therapy after an acute coronary syndrome: a systematic review and meta-analysis. Eur Heart J. 2013 Jun;34(22):1670-80. doi: 10.1093/eurheartj/eht049. Epub 2013 Mar 6. PMID 23470494
- [Background] Gibson CM, Mehran R, Bode C, Halperin J, Verheugt FW, Wildgoose P, Birmingham M, Ianus J, Burton P, van Eickels M, Korjian S, Daaboul Y, Lip GY, Cohen M, Husted S, Peterson ED, Fox KA. Prevention of Bleeding in Patients with Atrial Fibrillation Undergoing PCI. N Engl J Med. 2016 Dec 22;375(25):2423-2434. doi: 10.1056/NEJMoa1611594. Epub 2016 Nov 14. PMID 27959713
- [Background] Rubboli A, Saia F, Sciahbasi A, Bacchi-Reggiani ML, Steffanon L, Briguori C, Calabro P, Palmieri C, Rizzi A, Imperadore F, Sangiorgi GM, Valgimigli M, Carosio G, Steffenino G, Galvani M, Di Pasquale G, La Vecchia L, Maggioni AP, Bolognese L; WARfarin and Coronary STENTing (WAR-STENT) Study Group. Outcome of patients on oral anticoagulation undergoing coronary artery stenting: data from discharge to 12 months in the Warfarin and Coronary Stenting (WAR-STENT) Registry. J Invasive Cardiol. 2014 Nov;26(11):563-9. PMID 25363997
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Derived] Rigattieri S, Cristiano E, De Rosa S, Calabro P, Talarico GP, Cortese B, Caruso M, Redivo M, Musumeci G, Sciahbasi A. Peri-Procedural Management of Oral Anticoagulant Therapy in Patients Undergoing Percutaneous Coronary Intervention: Insights from the PERSEO Multicenter Registry. Catheter Cardiovasc Interv. 2025 Aug;106(2):1177-1186. doi: 10.1002/ccd.31657. Epub 2025 Jun 4. PMID 40468540
- [Derived] Sciahbasi A, De Rosa S, Gargiulo G, Giacoppo D, Calabro P, Talarico GP, Zilio F, Talanas G, Tebaldi M, Ando G, Rigattieri S, Misuraca L, Cortese B, Musuraca G, Lucci V, Guiducci V, Renda G, Zezza L, Versaci F, Giannico MB, Caruso M, Fischetti D, Colletta M, Santarelli A, Larosa C, Iannone A, Esposito G, Tarantini G, Musumeci G, Rubboli A. Management of Patients Treated With Oral Anticoagulant Therapy Undergoing Percutaneous Coronary Intervention With Stent Implantation: The PERSEO Registry. J Cardiovasc Pharmacol. 2024 Oct 1;84(4):457-467. doi: 10.1097/FJC.0000000000001607. PMID 39028879
- [Derived] Sciahbasi A, Gargiulo G, Talarico GP, Cesaro A, Zilio F, De Rosa S, Talanas G, Tebaldi M, Ando G, Rigattieri S, Misuraca L, Cortese B, Imperadore F, Lucci V, Guiducci V, Renda G, Zezza L, Versaci F, Giannico MB, Caruso M, Spaccarotella C, Calabro P, Esposito G, Tarantini G, Musumeci G, Rubboli A. Design of the PERSEO Registry on the management of patients treated with oral anticoagulants and coronary stent. J Cardiovasc Med (Hagerstown). 2022 Nov 1;23(11):738-743. doi: 10.2459/JCM.0000000000001372. Epub 2022 Sep 7. PMID 36166340

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03392948/Prot_SAP_000.pdf